CLINICAL TRIAL: NCT07005297
Title: Clinical Genetics Branch (CGB) Eligibility Screening Survey
Brief Title: Clinical Genetics Branch Eligibility Screening Survey
Status: Not yet recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002365; 002365-C
Record Dates: First submitted 2025-06-04; First posted 2025-06-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-09-19

CONDITIONS: Melanoma; Li-Fraumeni Syndrome; Pulmonary Blastoma; Chordoma; Congenital Bone Marrow Failure Syndromes; Costello Syndrome; Fanconi Anemia; CFC Syndrome (CFCS); Legius Syndrome; RASopathies
Keywords: Fanconi Anemia; Li-Fraumeni Syndrome; Clinical Genetics Branch, NCI; Hereditary Melanoma; Chordoma; DICER-1 syndrome; RASopathies; Cancer; Inherited Bone Marrow Failure Syndromes
MeSH Terms: conditions — Melanoma; Li-Fraumeni Syndrome; Pulmonary Blastoma; Chordoma; Congenital Bone Marrow Failure Syndromes; Costello Syndrome; Fanconi Anemia; Cardiofaciocutaneous syndrome; Legius syndrome; Melanoma, Cutaneous Malignant; Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: Prospective Cohort

SUMMARY:
Background:

Clinical Genetics Branch (CGB) researchers study individuals and populations at high genetic risk of cancer in order to improve our understanding of cancer and to improve cancer care. There are currently 6 open clinical genetics studies at the CGB eligible for this screening process.

* 02C0052: Etiologic Investigation of Cancer Susceptibility in Inherited Bone Marrow Failure Syndromes: A Natural History Study (Cancer in Bone Marrow Failure)
* 11C0255: Clinical, Epidemiologic, and Genetic Studies of Li-Fraumeni Syndrome (Li Fraumeni Syndrome Study)
* 11C0034: DICER1-Related Pleuropulmonary Blastoma Cancer Predisposition Syndrome: A Natural History Study (Pleuropulmonary Blastoma)
* 02C0211: Clinical, Laboratory, and Epidemiologic Characterization of Individuals and Families at High Risk of Melanoma (Melanoma-Prone Families)
* 10CN188: Genetic Clues to Chordoma Etiology: A Protocol to Identify Sporadic Chordoma Patients for Studies of Cancer-susceptibility Genes (Sporadic Chordoma Study)

The following studies have their own study-specific screeners. If you are interested in these studies, please click the links below to fill out the relevant study screener:

* 001109: Defining the Natural History of Squamous Cell Carcinoma in Fanconi anemia (SCC Screening in FA): https://service.cancer.gov/fanconi
* 20C0107: Clinical, Genetic, and Epidemiologic Study of Children and Adults with RASopathies (RASopathies Study): https://service.cancer.gov/myras

Objective:

To find people to participate in active CGB cancer research studies.

Eligibility:

People of any age who meet the eligibility criteria for one of the open CGB cancer research studies. You can learn more about the CGB cancer research studies by clicking on the links to the study-specific websites above. This typically involves a personal or family history of certain cancers that are being studied by researchers at CGB.

Design:

Participants will fill out a screening questionnaire to determine if they are eligible to participate in one or more CGB clinical genetics studies. The survey asks about personal health history, including cancer; family history; and genetic testing results and takes 15 to 20 minutes.

Each study has its own eligibility criteria. Survey respondents will select which study (or studies) that are interested in participating in, and the relevant study team(s) will review the screener to determine eligibility to participate in the study. Participants who are determined to be eligible for a study based on their screener will be contacted by the respective study team to learn more about the study and to consent to enroll in the study if they choose to do so. Participants who consent to enroll in a study may be asked to provide medical records; samples such as blood, saliva, or other tissues; and to participate in activities such as phone interviews or surveys. They may be invited for evaluations at the clinical center. Every study activity is voluntary. None of the studies provide treatments. Participants may be contacted to consider enrolling in future studies.

DETAILED DESCRIPTION:
Study Description:

This protocol will be utilized for the creation and management of an eligibility screening survey for patients who are interested in enrolling in a study being conducted by the Clinical Genetics Branch (CGB).

Objectives:

The primary objective of this protocol is to establish a database of eligibility data collected from prospective participants who have completed an eligibility screening survey. This database, managed by the CGB, will serve as a critical resource for assessing participant eligibility for enrollment in various CGB studies.

ELIGIBILITY:
* INCLUSION CRITERIA

There is no age restriction; therefore, viable neonates may be included. This eligibility screening protocol is intended for individuals meeting one or more of the following criteria:

1. Personal or family history of a diagnosis of a syndrome being actively investigated in one of the following CGB study protocol:

   * Protocol 000678: Medical history of neoplasia of an unusual type, pattern, or number.
   * Protocol 11C0255: A personal history of adrenal cortical carcinoma or choroid plexus carcinoma at any age, regardless of family history, or family or personal medical history of neoplasia consistent with the diagnosis of LFS or LFL.
   * Protocol 20C0107: Individuals with a clinical diagnosis of a RASopathy, including Costello syndrome, Noonan syndrome, Noonan syndrome with multiple lentigines, Cardiofaciocutaneous syndrome, Legius syndrome, capillary arteriovenous malformation syndrome, or others, are eligible. Published clinical diagnostic criteria exist for most of the clinical RASopathy syndromes and differ by syndrome. It will be uncommon for individuals to have a clinical diagnosis and not have had molecular genetic testing. All individuals considered by the study team to be at risk for a RASopathy who have not had prior genetic testing will have this completed as part of the study. The rare individuals with a clinical diagnosis of a RASopathy who are not found to carry a corresponding pathogenic or likely pathogenic variant in a known RASopathy gene will be considered for exome analysis for identification of potentially novel RASopathy germline variation.
   * Protocol 11C0034: An individual with histologically-confirmed PPB and/or other DICER1-related tumors
   * Protocol 02C0052: The participants will be affected by an IBMFS, or be members of a family with an IBMFS, and be at risk of being affected or carriers of the syndrome. Except for the rare X-linked recessive disorder (e.g. some dyskeratosis congenita patients), there should be equal numbers of male and female probands and family members. These IBMFS have been reported in most racial and ethnic groups, and thus all such groups will be included. The age range will be from birth to old age (grandparents of probands). The majority of the probands will be children (10-20% will be adults), and their parents and grandparents will be adults. All racial/ethnic groups are eligible.
   * Protocol 02C0211: Personal medical history of melanoma of an unusual type, pattern, or number diagnosed at any age.
   * Protocol 78C0039: Family or personal medical history of neoplasia of an unusual type, pattern, or number
2. Personal or family history of medical condition, malignancy, and/or benign neoplasm suggestive of hereditary cancer predisposition being actively investigated in the following CGB study protocol:

   * Protocol 000678: Known or suspected factor(s) predisposing to neoplasia, either genetic and/or congenital factors (birth defects, metabolic phenotype, chromosomal anomalies or Mendelian traits associated with tumors), environmental exposure (medications, occupation, radiation, diet, infectious agents, etc.), or unusual demographic features (very young age of onset, multiple tumors, etc.)
   * Protocol 11C0255: An individual with a sarcoma diagnosed under the age of 45; AND - At least one first-degree relative (parents, brothers, sisters and children) with a cancer of any kind diagnosed under the age of 45; AND - A third family member who is either a first- or second-degree relative (such as grandparents, aunts, uncles, nieces, nephews, and grandchildren) with cancer diagnosed under the age of 45 or having a sarcoma at any age.
   * Protocol 001109: On referral, persons >= 12 years with Fanconi Anemia (FA) primarily from North America will be included. An individual with FA who is 8 -11 years can also be included if they have a history of persistent oral potentially malignant lesion (OPMLs), dysphagia, or other concerning symptoms. Individuals with prior cancer diagnosis are eligible.
   * Protocol 11C0034: An individual from the general population with one or more of the unique tumors of the types associated with DICER1 including (but not exclusively), PPB, cystic nephroma, ovarian Sertoli-Leydig cell and other sex cordstromal tumors, ocular medulloepithelioma, nasal chondromesenchymal hamartoma, Wilms tumor, embryonal rhabdomyosarcoma, pineoblastoma, pituitary blastoma, ovarian sarcoma, CNS sarcoma and/or thyroid cancer - regardless of their family history. Additional DICER1-related neoplasms may be identified in the future, and they will be added to the protocol as needed
   * Protocol 02C0052: Fanconi anemia: FA patients have relatively specific birth defects, aplastic anemia, increased chromosome breakage in cells cultured with a DNA crosslinking agent such as mitomycin C (MMC) or diepoxybutane (DEB), pathogenic variant(s) in one of the cloned genes (six genes at this time), or assignment to one of the 7 or more complementation groups. Bone marrow failure is NOT required for the diagnosis, and approximately 25% do not have birth defects. FA has been diagnosed from birth to >50 years of age. FA Proven = positive chromosome breakage result, and/or pathogenic variant(s) in a known FANC gene. Patients in whom FA is suspected but whose chromosome breakage test is negative will still be considered if they have sufficient findings that lead the Principal Investigator to think they may be somatic mosaics and warrant further evaluation. Diamond Blackfan anemia: DBA patients have pure red cell aplasia with reticulocytopenia. Approximately 30% have physical abnormalities, often involving malformations of the thumbs. Approximately 90% are diagnosed within the first year of life. A pathogenic variant in a known DBA gene (RPS19 is currently the only known gene) is diagnostic, but lack of a pathogenic variant does not rule out DBA, since the cloned gene is responsible for only approximately 25% of the disease. Since many cases are sporadic or occur in families with silent carriers, patients without a positive family history will be included. Currently DBA is diagnosed by clinical findings after exclusion of known causes of red cell aplasia. Approximately 90% have elevated red cell adenosine deaminase levels, a finding which is supportive, but not diagnostic, of DBA. Dyskeratosis congenita: DC patients develop dyskeratotic nails, lacy hyperpigmentation of the skin and mucous membrane leukoplakia as they age (the diagnostic clinical triad; two of the three are required for a firm diagnosis). Findings in young patients may be very subtle, and diagnoses are usually made in teenagers or young adults. More than 75% are male. DC patients are often diagnosed without hematologic abnormalities by dermatologists; however, some patients present with aplastic anemia prior to the evolution of the syndrome-related physical features. A pathogenic variant in the DKC1 gene is diagnostic, but normal DKC1 does not exclude DC. The diagnosis is often clinical, after exclusion of FA and other IBMFS. Shwachman Diamond Syndrome: SDS patients have neutropenia, malabsorption and failure to thrive due to exocrine pancreatic insufficiency. The gene has not yet been cloned. Pancreatic insufficiency is documented by direct measurement of pancreatic enzymes, low serum immunoreactive trypsinogen, or elevated fecal fat levels. Neutropenia requires an absolute neutrophil count of <1500/mm3 on multiple occasions. Other causes of malabsorption such as cystic fibrosis, Pearson syndrome, and Johansson-Blizzard syndrome must be excluded. Cystic fibrosis will be excluded in patients who have a positive sweat test performed at an approved CF center. Amegakaryocytic thrombocytopenia: These patients have early onset thrombocytopenia (<150,000/mm3), usually within the first year of life, due to absent, diminished, or abnormal bone marrow megakaryocytes, without antiplatelet antibodies. Physical examination is often normal; in particular, there are no abnormalities of the radial rays. Pathogenic variant(s) in the MPL gene are diagnostic, but normal MPL does not exclude this diagnosis. Thrombocytopenia absent radii: TAR patients have absent radii, usually bilateral, with intact thumbs (in contrast with FA and trisomy 18, where thumbs are absent if radii are absent), and thrombocytopenia at birth. Other radial aplasia syndromes such as Holt-Oram syndrome or VATER syndrome must be excluded. Severe Congenital Neutropenia: Patients with SCN have persistent and noncyclic low absolute neutrophil counts, with more than 2 measurements <200/mm3, and a history of pyogenic infections during the first year of life, and bone marrow maturation arrest at the promyelocyte/myelocyte stage. They do not have birth defects, and they usually have normal hemoglobin and platelet counts. They are designated Kostmann Syndrome (KS) only if there is a pattern of autosomal recessive inheritance. Pathogenic variant(s) in the neutrophil elastase gene (ELA2) are supportive of the diagnosis of SCN, but do not distinguish SCN patients from those with cyclic neutropenia, which is milder and not preleukemic. Many of the cases of SCN have been shown to be due to dominant pathogenic variant(s)s in ELA2. Pearson Syndrome: Pearson syndrome consists of malabsorption, neutropenia, alone or with anemia and/or thrombocytopenia, and metabolic acidosis. Onset is in infancy or early childhood. The diagnosis is strongly suspected if bone marrow examination reveals vacuoles in myeloid and erythroid progenitors, and ring sideroblasts. Confirmation derives from detection of deletions in mitochondrial DNA, which range from 2 to 8 kb in size, and include the respiratory enzymes. Absence of reports to date of cancer or leukemia in this syndrome may derive from early death due to the metabolic problems. Other bone marrow failure syndromes: There are occasional patients with a pattern of hematologic abnormalities, physical findings, malignancies, or family histories which are not characteristic of the syndromes described above, but which nonetheless suggests that they have a genetic bone marrow failure syndrome. There may be similar cases in the literature, or in the experience of the investigator, which may ultimately lead to assignment of these patients to a known or new syndrome. There are additional bone marrow failure syndromes which are even more rare, such as Revesz, WT, IVIC, radio-ulnar synostosis, ataxia-pancytopenia, etc. Syndromic classification of extremely rare disorders is facilitated if they are collected in one center. Since malignancy is often part of these syndromes, they will be eligible for enrollment in this protocol.
   * Protocol 02C0211: Known or suspected factor(s) predisposing to melanoma, either genetic or congenital factors (giant congenital nevi, dysplastic nevi, Spitzoid tumors), or unusual demographic features (e.g., very young age of onset, multiple melanomas, previous history of heritable retinoblastoma, Hodgkin's disease, lymphoma, immunodeficiency syndrome, or organ transplant).
   * Protocol 10CN188: Diagnose with chordoma or related tumor at any age and any primary site.
   * Protocol 78C0039: Known or suspected factor(s) predisposing to neoplasia, either genetic and/or congenital factors (birth defects, metabolic phenotype, chromosomal anomalies or Mendelian traits associated with tumors), environmental exposure (medications, occupation, radiation, diet, infectious agents, etc.), or unusual demographic features (very young age of onset, multiple tumors, etc.). Personal and family medical history must be verified through questionnaires, interviews, and review of pathology slides and medical records. For familial neoplasms, two or more living affected cases among family members are required. The types of familial tumors that we are currently actively accruing include Familial Cancers: bladder, brain, chordoma, lung, nevoid basal cell carcinoma syndrome (NBCC) Familial Benign Neoplasms: meningiomas, neurofibromatosis 2 (bilateral acoustic neurofibromatosis) The types of familial tumors under active accrual and study are predominantly investigator- and hypothesis-driven. This approach permits CGB investigators to remain alert to the opportunities afforded by clusters of rare tumors in families and individuals, and to be more responsive to the dynamic research priorities in cancer genetics.
3. Personal or family history of a genetic variant in a hereditary cancer predisposition being actively investigated in the following CGB study protocols:

   * Protocol 11C0255: A personal history of a germline TP53 mutation; or, - A first or second- degree relative of a TP53 mutation carrier, regardless of mutation status
   * Protocol 20C0107: Individuals with a germline variant (P/LP or a variant of uncertain significance but predicted bioinformatically to be damaging) in a RASopathy-associated gene are eligible. These include but are not limited to: BRAF, CBL, HRAS, KRAS, LZTR1, MAP2K1, MAP2K2, MAP3K8, MRAS, NRAS, PPP1CB, PTPN11, RAF1, RASA1, RASA2, RIT1, RRAS, SHOC2, SOS1, SPRED1. From herein, we refer to 1) individuals with germline pathogenic variation in a RAS pathway gene AND 2) individuals with a clinical RASopathy diagnosis but in whom a genetic variant has not yet been identified as "carriers." The first member of a family to be identified is termed a "proband."
   * Protocol 11C0034: An individual with a known or suspected DICER1 disease associated variant.
   * Protocol 02C0052: An individual with a pathogenic variant(s) in a known FANC gene. Individual with Diamond Blackfan Anemia with a pathogenic variant in a known DBA gene (RPS19). Individuals with Dyskeratosis congenita with a pathogenic variant in the DKC1 gene. Individuals with Amegakaryocytic thrombocytopenia with pathogenic variants) in the MPL gene. Individuals with Severe Congenital Neutropenia with a pathogenic variant(s) in the neutrophil elastase gene (ELA2).

EXCLUSION CRITERIA

While this protocol is intended to be used by those meeting the inclusion criteria above, there are no explicit exclusion criteria for this study, since the initiative to complete the eligibility screener survey is at the will of the participant or his or her parent/guardian/LAR.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People of any age who meet the eligibility criteria for one of the open CGB cancer research studies. This typically involves a personal or family history of certain cancers that are being studied by researchers at CGB.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2035-01-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Eligible Participants Identified | Duration of the protocol
  The total count of individuals who qualify for a CGB study

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Savage, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No